CLINICAL TRIAL: NCT07170982
Title: A Randomized, Controlled, Multicenter Clinical Study of Fruquintinib Combined With Standard Chemotherapy Versus Standard Chemotherapy as First-line Treatment for Advanced pMMR Endometrial Cancer
Brief Title: Fruquintinib Combined With Standard Chemotherapy Versus Standard Chemotherapy as First-line Treatment for Advanced pMMR Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jihong Liu, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-E001
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm/Group 1 (Experimental): Trial Group: Fruquintinib + standard chemotherapy (trial drug includes fruquintinib);
  * Fruquintinib: The recommended dose is based on the results of the safety run-in phase: once daily, orally, on days 1-14, every 3 weeks, on an empty stomach or after a meal, preferably with 100-200 ml of drinking water.
  * Paclitaxel: 175 mg/m², IV drip, day 1, every 3 weeks, intravenous infusion over at least 3 hours;
  * Carboplatin: Area under the plasma concentration-time curve (AUC) 5 mg/mL/min, IV drip, day 1, every 3 weeks, intravenous infusion over at least 1 hour.
  During the study, it is recommended that carboplatin be administered after the completion of the paclitaxel infusion, or according to local clinical practice.
  Interventions: Drug: Fruquintinib
- Arm/Group 2 (No Intervention): Control group: Standard chemotherapy regimen (paclitaxel + carboplatin);
  * Paclitaxel: 175 mg/m², iv drip, day 1, every 3 weeks, intravenous infusion for at least 3 hours;
  * Carboplatin: Area under the plasma concentration-time curve (AUC) 5 mg/mL/min, iv drip, day 1, every 3 weeks, intravenous infusion for at least 1 hour.

INTERVENTIONS:
Drug: Fruquintinib — This study aims to confirm the safety and efficacy of fruquintinib combined with standard chemotherapy, further compare whether first-line standard chemotherapy has superiority, bring better survival benefits to patients with pMMR endometrial cancer, and provide more options for patients with late recurrent and metastatic endometrial cancer.
  Arms: Arm/Group 1

SUMMARY:
This is a randomized, controlled, multicenter clinical study designed to explore the safety and efficacy of fruquintinib combined with standard chemotherapy versus standard chemotherapy as first-line treatment for advanced mismatch repair-intact (pMMR) endometrial cancer. The standard chemotherapy regimen is TC (paclitaxel + carboplatin);

Safety introduction period (N=12):

Dose expansion phase (N=116): Subjects who met the inclusion criteria were randomly assigned 1:1 to the following treatment groups:

Experimental group: fruquintinib + standard chemotherapy (trial drugs include fruquintinib); Control group: standard chemotherapy TC regimen (paclitaxel + carboplatin); The study treatment cycle was 21 days, with a maximum of 6 cycles of paclitaxel and carboplatin. Patients who achieved disease control or better entered the maintenance treatment phase. The experimental group received maintenance treatment with fruquintinib monotherapy until one of the following conditions occurred: PD (except for cases where continued treatment after PD was allowed as stipulated in the protocol), death, intolerable toxicity, or other criteria for termination of study treatment stipulated in the protocol, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must voluntarily participate in the study, sign the informed consent form, and demonstrate good compliance; 2. Age 18-75 years (inclusive); 3. Body mass index (BMI) ≥18.5 kg/m²; 4. Histologically or cytologically confirmed stage III/IV or recurrent/metastatic endometrial cancer with measurable or evaluable lesions as assessed by the investigator according to RECIST 1.1 (excluding lesions in cavitary organs (e.g., vagina); if the only measurable or evaluable lesion is a lesion previously treated with local therapy (radiotherapy, ablation, vascular intervention, etc.), there must be clear radiographic evidence of PD in that lesion; 5. No prior first-line systemic anticancer therapy (patients with recurrence after 6 months of adjuvant or neoadjuvant therapy are permitted); 6. Immunohistochemistry results demonstrating pMMR; 7. ECOG performance status 0-1; 8. Expected survival ≥ 6 months; 9. Adequate bone marrow, liver, and kidney function;

  1. Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L, platelets ≥100 × 10⁹/L, and hemoglobin ≥90 g/L (no blood transfusion or blood product use within 14 days prior to the laboratory test, and no granulocyte colony-stimulating factor or other hematopoietic stimulating factor use within 7 days prior to the laboratory test);
  2. Serum total bilirubin ≤1.5 times the upper limit of normal (ULN);
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN in the absence of liver metastasis; ALT and AST ≤5 × ULN in the presence of liver metastasis;
  4. Serum creatinine ≤1.5 × ULN and creatinine clearance ≥50 mL/min;
  5. Urinalysis shows urine protein <2+; if urine protein ≥2+, the 24-hour urine protein count should be <1 g;
  6. International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

     10. Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to treatment and be willing to use medically approved effective contraception (e.g., intrauterine device, contraceptive device, or condom) during the study and for 6 months after the last dose of study drug; or be advised to use effective contraception during the study and for 3 months after the last dose of study drug.

     Exclusion Criteria:
* 1. Endometrial sarcoma; 2. Receipt of approved systemic anti-cancer therapy within 4 weeks prior to enrollment, including chemotherapy, biological therapy, targeted therapy, hormone therapy, or traditional Chinese medicine (for traditional Chinese medicine treatments with clear anti-cancer indications in the package insert, a one-week washout period prior to enrollment is sufficient); 3. Other malignancies within the past 5 years (excluding cured basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix); 4. Central nervous system (CNS) metastases in the past or during the screening period; 5. Radical radiotherapy (including more than 25% bone marrow radiotherapy) within 4 weeks prior to enrollment; brachytherapy (e.g., implantation of radioactive particles) within 60 days prior to enrollment; or palliative radiotherapy for bone metastases within 1 week prior to enrollment; 6. Previous treatment with any anti-programmed death receptor 1 (PD-1), anti-PD-L1, anti-PD-L2, or anti-cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibody, or any other antibody targeting T cell co-stimulation or checkpoint pathways (e.g., OX40, CD137, etc.), or small molecule vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitors; 7. Use of immunosuppressants within 4 weeks prior to enrollment, excluding topical glucocorticoids administered by nasal spray, inhalation, or other routes, or physiological doses of systemic glucocorticoids (i.e., no more than 10 mg/day of prednisone or equivalent doses of other glucocorticoids). Temporary use of glucocorticoids for dyspnea due to conditions such as asthma and chronic obstructive pulmonary disease is permitted, as is the use of prophylactic corticosteroids to prevent allergic reactions (e.g., pretreatment before administration of intravenous contrast agents or chemotherapy drugs); 8. Any active autoimmune disease requiring systemic treatment or a history of an autoimmune disease within the past two years, including but not limited to uveitis, inflammatory bowel disease, hepatitis, hypophysitis, vasculitis, systemic lupus erythematosus, etc. (Patients with vitiligo, psoriasis, alopecia, or Grave's disease who have not required systemic treatment within the past two years and type 1 diabetes requiring only insulin replacement therapy are eligible); a known history of primary immunodeficiency; patients with only positive autoimmune antibodies must have the presence of an autoimmune disease confirmed at the investigator's discretion.

  9. Major surgery within four weeks prior to enrollment (the definition of major surgery is based on Level 3 and Level 4 surgery as defined in the "Regulations on the Administration of Clinical Application of Medical Technology," effective May 1, 2009) or unhealed wounds or fractures assessed by the investigator as clinically significant; or anticipated need for major surgery during the study (excluding diagnostic procedures); fistula formation must be stable for four weeks. Tissue aspiration or endoscopic biopsy within seven days prior to enrollment is excluded. Note: Implantation of a central venous access catheter (e.g., an infusion port or similar device) is permitted.

  10. Uncontrolled malignant pleural effusion, ascites, or pericardial effusion (defined as ineffectively controlled by diuretics or paracentesis, as determined by the investigator); 11. Patients currently have uncontrolled hypertension, defined as: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg; 12. Patients currently have any disease or condition that affects drug absorption, or patients are unable to take oral medications; 13. Patients currently have active, large, or deep gastric or duodenal ulcers, ulcerative colitis, or other gastrointestinal diseases with active bleeding from unresected tumors, or severe gastrointestinal disorders (infection, obstruction, diarrhea ≥ Grade 1, etc.), or other conditions determined by the investigator to be potentially causing gastrointestinal bleeding or perforation; or gastrointestinal perforation or gastrointestinal fistula that has not resolved after surgical treatment; 14. Arterial thrombosis or deep vein thrombosis within 6 months prior to enrollment; or stroke and/or transient ischemic attack within 12 months; thrombosis caused by an implantable intravenous infusion pump or catheter, excluding those whose thrombosis has stabilized after conventional anticoagulation.

  15. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months prior to enrollment; congestive heart failure New York Heart Association (NYHA) class 2 or higher; left ventricular ejection fraction (LVEF) <50%; known history of aneurysm.

  16. Active infection or unexplained fever (temperature >38.5°C) prior to enrollment.

  17. Patients with active pulmonary tuberculosis (TB) who are currently receiving anti-TB treatment or have received anti-TB treatment within 1 year prior to enrollment.

  18. Patients with a history or current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, or severe lung function impairment that may interfere with the detection and management of suspected drug-related pulmonary toxicity; patients with a history or current history of (non-infectious) lung inflammation requiring steroid therapy; 19. Positive human immunodeficiency virus (HIV) antibody screening; 20. Known history of clinically significant liver disease, including active viral hepatitis infection [positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) with hepatitis B virus deoxyribonucleic acid (HBV DNA) > 1 × 104 copies/mL or > 2000 IU/mL; known positive hepatitis C virus antibody (HCV Ab) with HCV RNA > 1 × 103 copies/mL], other hepatitis, or clinically significant moderate to severe cirrhosis; 21. Known hypersensitivity to any study drug (fruquintinib, paclitaxel, or carboplatin) or any of its excipients, or a history of severe allergic reaction to any other monoclonal antibody; 22. Receipt of other clinical medications not approved or marketed in China within 4 weeks prior to enrollment; 23. Patients with known psychiatric illness or substance abuse disorder that may affect study compliance; 24. Patients deemed by the investigator to be unsuitable for participation in this clinical study for other reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 years
  It refers to the proportion of patients whose tumor shrinks to a certain amount and remains so for a certain period of time, including cases of CR and PR.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  PFS is defined as the time from the date of treatment receipt to the first occurrence of disease progression or death from any cause, whichever occurs first. The Kaplan-Meier method was used to estimate PFS and calculate the 95% confidence interval.
Disease control rate (DCR) | 3 years
  The percentage of patients who achieved confirmed complete response (CR), partial response (PR), and stable disease (SD) among those who could be evaluated for efficacy.
Time to response (TTR) | 3 years
  The time from randomization to the earliest CR or PR (whichever occurs first) is calculated only for patients with a BOR of CR or PR.
Overall survival (OS) | 4 years
  OS refers to the period from enrollment to death from any cause. For subjects still alive at the last follow-up, OS was censored based on the last follow-up date. The analysis method was the same as for PFS.
AE | 4 years
  Adverse events
HRQoL | 3 years
  Health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Ph. D, Principal Investigator — Sun Yat-sen University Cancer
Locations (1):
- Department of Gynecologic Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China